CLINICAL TRIAL: NCT06141590
Title: A Clinical Study to Evaluate the Safety and the Pharmacokinetics of UI068 in Healthy Adult Volunteers Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea United Pharm. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KUP-UI068-101
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UI068 (Experimental)
  Interventions: Drug: administration of UI068
- UIC202205, UIC202206 (Experimental)
  Interventions: Drug: administration of UIC202205, UIC202206

INTERVENTIONS:
Drug: administration of UI068 — Test
  Arms: UI068
Drug: administration of UIC202205, UIC202206 — Reference
  Arms: UIC202205, UIC202206

SUMMARY:
This study was open-label, randomized, fed, single-dose, 2-groups, 2 periods, crossover designe to compare the safety and pharmacokinetics of UI068 and co-administration of UIC202205 and UIC202206.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects over the ages of 19 at screening
* Subjects whose body weight over 60 kg and having a body mass index (BMI) of over than 18.0 and less than 30.0 kg/m2 at screening (☞ BMI(kg/m2) = Weight(kg)/{Height(m)}2)
* There are no clinically significant congenital diseases/chronic diseases/ pathological symptoms or finding at the screening
* he principal investigator determines to be suitable test subjects as a result of diagnostic tests and electrocardiogram tests etc.
* From the date of first to the last administration of the investigational drug Until 7 weeks , tester or spouse or partner must use a method of contraception recognized in clinical trials.
* The tester who is signed after being explained and understanding about purpose and content of this clinical trial, characteristics of the investigational drug.

Exclusion Criteria:

* Clinically significant diseases related to the digestive system, cardiovascular system, endocrine system, respiratory system, blood/tumor, infectious disease, kidney and genitourinary system, mental/nervous system, musculoskeletal system, immune system, ENT system, skin system, and ophthalmic system. Those who have or have a history of
* Those with a history of gastrointestinal surgery (excluding simple appendectomy or hernia surgery) that may affect drug absorption or gastrointestinal disease
* Those who took drugs that induce or inhibit drug-metabolizing enzymes, such as barbiturates, within 1 month of the first dose, or took drugs that may interfere with this clinical trial within 10 days of the first dose.
* A person who participated in another clinical trial or bioequivalence test and administered an investigational drug within 6 months of the first administration date
* Those who donated whole blood or component blood within 2 weeks or received a blood transfusion within 4 weeks of the first administration date
* Those who meet the following conditions within 1 month of the first medication date

  * Alcohol consumption exceeding 21 drinks/week on average for men
  * For women, alcohol consumption exceeds an average of 14 drinks/week

    (1 glass = 50 mL of soju or 30 mL of liquor or 250 mL of beer)
  * Smoking more than 20 cigarettes per day on average
* Those who fall under the following

  * Patients with hypersensitivity to clinical investigational drugs or ingredients contained in clinical investigational drugs
  * Persons with a history of hypersensitivity to biguanide drugs
* Patients with the following diseases

  * Patients with moderate (stage3b) and severe renal impairment (eGFR<45mL/min/1.73m2), Acute conditions that can affect kidney function, such as diabetes, serious infections, cardiovascular collapse (shock), acute myocardial infarction, and sepsis
  * Patients with acute and unstable heart failure
  * Patients undergoing tests requiring intravenous administration of radioiodine contrast material (e.g., intravenous urography, intravenous cholangiography, angiography, computed tomography using contrast agent, etc.)
  * Patients with acute or chronic metabolic acidosis, including type 1 diabetes, lactic acidosis, diabetic ketoacidosis with or without coma, and patients with a history of ketoacidosis
  * Diabetic precoma
  * Patients with severe infections or severe traumatic systemic disorders
  * Patients with malnutrition, starvation, weakness, pituitary dysfunction or adrenal dysfunction
  * Patients with acute or chronic diseases that can cause tissue hypoxia such as liver dysfunction, respiratory failure, acute myocardial infarction, and shock, excessive alcohol intake, and gastrointestinal disorders such as dehydration, diarrhea, and vomiting
* Persons judged by the principal investigator to be unsuitable for participation in this clinical trial for reasons other than the above selection/exclusion criteria
* For female volunteers, those who are pregnant, suspected of being pregnant, or lactating

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-03-11 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
AUCt | 0 to 72hr
  Evaluation PK for Linagliptin and Metformin after single dose
Cmax | 0 to 72hr
  Evaluation PK for Linagliptin and Metformin after single dose

CONTACTS AND LOCATIONS:
Locations (1):
- H plus Yangji Hospital, Seoul, Gwanak-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided